CLINICAL TRIAL: NCT05769946
Title: A Phase II Study to Evaluate the Efficacy and Safety of Hemay005 Tablet in Adult With Moderate to Severe Atopic Dermatitis
Brief Title: A Study of Hemay005 in Adult With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM005AD2S01
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Hemay005, Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Hemay005

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- placebo (Placebo Comparator): Atopic dermatitis patients treated with placebo for 12 week.
  Interventions: Drug: Hemay005
- Hemay005 60mg (Experimental): Atopic dermatitis patients treated with Hemay005 60mg BID for 12 week.
  Interventions: Drug: Hemay005
- Hemay006 75mg (Experimental): Atopic dermatitis patients treated with Hemay005 75mg BID for 12 week.
  Interventions: Drug: Hemay005

INTERVENTIONS:
Drug: Hemay005 — A PDE-4 inhibitor

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled, phase II study to evaluate the efficacy and safety of Hemay005 tablet in the treatment of moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign the informed consent form for this study;
* 18-75 years old (including boundary value) , gender is not limited;
* Ability to adhere to follow-up schedules and other program requirements;
* According to Hanifin & Rajka diagnostic criteria of atopic dermatitis (AD) , the patients with AD history ≥6 months;
* At baseline, the severity of AD was moderate to severe: IGA score was 3 or more, and the area of involved skin lesion was 10% BSA or more;
* Participants were required to use contraception during the study period.

Exclusion Criteria:

* A medical history unsuitable for participation in a clinical study；
* Pregnant or lactating women；
* Allergic to the drug or its preparation；
* Patients who had undergone major surgery within 6 months before screening or who were scheduled for major surgery during the trial period；
* Participants who had participated in any drug or device clinical trial within the previous 3 months were screened；
* Vaccination with live or attenuated vaccines is planned for the duration of the trial；
* Any drugs is taking that may affect the effectiveness evaluation;
* Any clinically significant abnormality in 12-lead ECG at screening that was judged by the investigator as unsuitable for inclusion；
* When investgater believe that any condition could lead to unnecessary risks for patients participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
EASI-75 | week 12
  Percentage of subjects reaching 75% or higher improvement from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No